CLINICAL TRIAL: NCT03272477
Title: A Prospective, Randomized, Multicenter, Open-label Comparison of Pre-surgical Combination of Trastuzumab and Pertuzumab With Concurrent Taxane Chemotherapy or Endocrine Therapy Given for Twelve Weeks With a Quality of Life Assessment of Trastuzumab, Pertuzumab in Combination With Standard (Neo)Adjuvant Treatment in Patients With Operable HER2+/HR+ Breast Cancer.
Brief Title: Study to Compare Neoadjuvant Combination of Trastuzumab and Pertuzumab With Concurrent Taxane Chemotherapy or Endocrine Therapy and Quality of Life Assessment Under Adjuvant Therapy in Operable HER2+/HR+ Breast Cancer Patients
Acronym: TP-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palleos Healthcare GmbH (Industry)
Collaborators: Roche Pharma AG (Industry); WSG WOMEN´S HEALTHCARE STUDY GROUP (Unknown); Cankado GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH002-TP-II
Record Dates: First submitted 2017-08-10; First posted 2017-09-05 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Breast Neoplasms
Keywords: hormone receptor positive; human epidermal growth factor receptor 2 positive; Early breast cancer; HR+/HER2+
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Tamoxifen; Paclitaxel; Epirubicin; Cyclophosphamide; Anastrozole; Letrozole; exemestane; Leuprolide; Goserelin; Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel+Trastuzumab+Pertuzumab (Active Comparator): Neoadjuvant therapy: Trastuzumab and Pertuzumab in a 3-weekly schedule in combination with standard Taxane chemotherapy.
  Adjuvant Therapy: Standard of care
  Interventions: Drug: Perjeta Injectable Product; Drug: Herceptin; Drug: Tamoxifen; Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Leuprorelin acetate; Drug: Goserelin; Diagnostic Test: Biopsy; Procedure: Surgery
- Endocrine+Trastuzumab+Pertuzumab (Experimental): Neoadjuvant therapy: Trastuzumab and Pertuzumab in a 3-weekly schedule in combination with endocrine therapy.
  Adjuvant Therapy: Standard of care
  Interventions: Drug: Perjeta Injectable Product; Drug: Herceptin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Paclitaxel; Drug: Tamoxifen; Drug: Leuporelin acetate; Drug: Goserelin; Diagnostic Test: Biopsy; Procedure: Surgery

INTERVENTIONS:
Drug: Perjeta Injectable Product — Single dose of 840mg (loading dose) day1 cycle 1, 420mg at day1 of each subsequent cycle, every 3 weeks. (The latter cycle is called cycle of treatment and is to be given 4 times in the neoadjuvant phase and 14 times in the adjuvant therapy phase.)
  Other Names: Pertuzumab
Drug: Herceptin — Single dose of 8mg/kg (loading dose) day1 cycle 1; 6mg/kg at day1 of each subsequent cycle body weight every 3 weeks. (This is called cycle of treatment and is to be given four times in the neoadjuvant phase and 14 times in the adjuvant therapy phase.)
  Other Names: Trastuzumab
Drug: Tamoxifen — 20 mg per day for a total of 40 weeks in the adjuvant therapy phase.
  Arms: Paclitaxel+Trastuzumab+Pertuzumab
Drug: Paclitaxel — 80mg/sqm, day one of each cycle, every week. This is called a cycle of treatment and is to be given for 12 weeks in neoadjuvant therapy phase.
  Arms: Paclitaxel+Trastuzumab+Pertuzumab
Drug: Epirubicin — 12 weeks (4cycles) of max. 90mg/sqm in adjuvant therapy phase
Drug: Cyclophosphamide — 12 weeks (4cycles) of 600 mg/sqm i.v. on day 1+8 or 12 weeks (4cycles) of 500 mg/sqm i.v. on day 1 in adjuvant therapy phase
Drug: Anastrozole — 1mg per day for a total of 40 weeks in adjuvant therapy phase
  Arms: Paclitaxel+Trastuzumab+Pertuzumab
Drug: Letrozole — 2,5 mg/day for a total of 40 weeks in adjuvant therapy phase
  Arms: Paclitaxel+Trastuzumab+Pertuzumab
Drug: Exemestane — 25mg/day for a total of 40 weeks in adjuvant therapy phase
  Arms: Paclitaxel+Trastuzumab+Pertuzumab
Drug: Leuprorelin acetate — One injection of 3,75mg every month or 4 weeks in pre-menopausal women treated with aromatase inhibitors Anastrozole or Letrozole or Exemestane, for a total of 40 weeks in the adjuvant therapy phase.
  Arms: Paclitaxel+Trastuzumab+Pertuzumab
Drug: Goserelin — 3,6mg every 28 days or 4 weeks in pre-menopausal women treated with aromatase inhibitors Anastrozole or Letrozole or Exemestane, for a total of 40 weeks in the adjuvant therapy phase.
  Arms: Paclitaxel+Trastuzumab+Pertuzumab
Drug: Anastrozole — 1mg per day for 12 weeks in neoadjuvant therapy phase; 1mg per day for a total of 40 weeks max. in adjuvant therapy phase
  Arms: Endocrine+Trastuzumab+Pertuzumab
Drug: Letrozole — 2,5 mg per day for 12 weeks in neoadjuvant therapy phase; 2,5 mg perday for a total of 40 weeks max. in adjuvant therapy phase
  Arms: Endocrine+Trastuzumab+Pertuzumab
Drug: Exemestane — 25mg/day for 12 weeks in neoadjuvant therapy phase; 25mg/day for a total of 40 weeks max. in adjuvant therapy phase
  Arms: Endocrine+Trastuzumab+Pertuzumab
Drug: Paclitaxel — 80mg/sqm, day one of each cycle, every week. This is called a cycle of treatment an is to be given for 12 weeks in the adjuvant phase
  Arms: Endocrine+Trastuzumab+Pertuzumab
Drug: Tamoxifen — 20mg per day (given over 12 weeks in the neoadjuvant therapy phase and over 40 weeks max. in the adjuvant therapy phase.
  Arms: Endocrine+Trastuzumab+Pertuzumab
Drug: Leuporelin acetate — One injection of 3,75mg every month or 4 weeks in pre-menopausal women treated with aromatase inhibitors Anastrozole or Letrozole or Exemestane (given over 12 weeks in the neoadjuvant therapy phase and over 40 weeks max. in the adjuvant therapy phase).
  Arms: Endocrine+Trastuzumab+Pertuzumab
Drug: Goserelin — 3,5mg every 28 days or 4 weeks in pre-menopausal women treated with aromatase inhibitors Anastrozole or Letrozole or Exemestane (given over 12 weeks in the neoadjuvant therapy phase and over 40 weeks max. in the adjuvant therapy phase).
  Arms: Endocrine+Trastuzumab+Pertuzumab
Diagnostic Test: Biopsy — Core biopsy at screening (outside of protocol), at week 4 after randomization, (at week 14 in addition if neoadjuvant phase is prolonged)
Procedure: Surgery — Surgery at week 14 after randomization (or later, if neoadjuvant phase is prolonged)

SUMMARY:
This is a prospective, phase IIa, multicenter, randomized, open-label study comparing a pre-surgical combination of trastuzumab and pertuzumab with concurrent weekly paclitaxel chemotherapy or endocrine therapy given for 12 weeks with a quality of life assessment for 40 additional weeks in patients with operable HER2+/HR+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age at diagnosis 18 years and older
* Histologically confirmed unilateral primary invasive carcinoma of the breast
* Patients must qualify for neoadjuvant treatment as follows:

  * No clinical evidence for distant metastasis (M0)
  * Clinical cT1c-T4a-c (participation of patients with tumors > cT2 is strongly recommended) and no evidence for distant metastases (M0)
  * All clinical N (participation of patients with cN+, also in case of cT1c, is strongly recommended)
  * Known positive HR-status and centrally confirmed HER2+-status by IHC/FISH
  * Patients need to fulfill adequate blood count and organ function to receive chemotherapy (see exclusion criteria).
* Tumor block available for central pathology review
* Performance Status ECOG ≤ 1 or KI ≥ 80%
* Negative pregnancy test (urine or serum) within 7 days prior to registration in premenopausal patients
* Patients of childbearing potential must accept to implement a highly effective (less than 1% failure rate according to Pearl index) non-hormonal contraceptive measures during the study treatment and for 6 months following the last dose of study treatment (trastuzumab and pertuzumab) such as:

  * Intrauterine device (IUD)
  * bilateral tubal occlusion
  * vasectomised partner
  * sexual abstinence
* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
* The patient must be accessible for treatment and follow-up
* LVEF > 55%; LVEF within normal limits of each institution measured by echocardiography (within 42 days prior to randomization)
* Normal ECG (within 42 days prior to randomization)

Exclusion Criteria:

* Known hypersensitivity reaction to the compounds or incorporated substances
* Prior malignancy with a disease-free survival of < 10 years, except curatively treated basalioma of the skin, pTis of the cervix uteri
* Non-operable breast cancer including inflammatory breast cancer
* Previous or concurrent treatment with cytotoxic agents for any reason
* Concurrent treatment with other experimental drugs and participation in another clinical trial or clinical research project within 30 days prior to study entry is excluded
* Male breast cancer
* Concurrent pregnancy
* Breastfeeding
* Sequential breast cancer
* Reasons indicating risk of poor compliance
* Known polyneuropathy ≥ grade 2
* Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study including but not confined to:

  * Uncompensated chronic heart failure or systolic dysfunction (LVEF < 55%, CHF NYHA classes II-IV),
  * unstable arrhythmias requiring treatment i.e., atrial tachycardia with a heart rate ≥ 100/min at rest, significant ventricular arrhythmia (ventricular tachycardia) or higher-grade AV-block,
  * Angina pectoris within the last 6 months requiring anti-anginal medication,
  * Clinically significant valvular heart disease,
  * Evidence of myocardial infarction on electrocardiogram (ECG),
  * Poorly controlled hypertension (e.g., systolic > 180 mm Hg or diastolic > 100 mm Hg).
* Inadequate organ function including but not confined to:

  * hepatic impairment (Child Pugh Class C)
  * pulmonary disease (severe dyspnea at rest requiring oxygen therapy)
* Abnormal blood values:

  * Thrombocytopenia > CTCAE grade 1
  * Increases in ALT/AST > CTCAE grade 1
  * Hypokalaemia > CTCAE grade 1
  * Neutropenia > CTCAE grade 1
  * Anaemia > CTCAE grade 1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 14 weeks after start of therapy treatment
  14 weeks after start of therapy treatment, tumor and lymph node biopsy is performed to reach the primary endpoint of pathological complete response (pCR) which is defined as the absence of residual invasive cancer of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (ypT0/is ypN0 in the current AJCC staging system). As secondary endpoint, also other response states will be taken into account: no invasive tumor in the complete resected breast specimen irrespective of the lymph node state following completion of neoadjuvant systemic therapy (ypT0/is, any ypN).

SECONDARY OUTCOMES:
Health-related quality of life using EORTC QBL-BR-23 scale | During the neoadjuvant treatment phase at baseline (week 1) and at week 13. In the adjuvant therapy phase, every 3 month, up to 12 months (from date of randomization) or date of drop out, whatever comes first
  Assessment of quality of life questions during the past week or during the past 4 weeks (depending on the questions) are measured on a 4 level-scale: 1 (not at all); 2 (a little); 3 (quite a bit); 4 (very much)
Health-related quality of life using EQ5D-5L scale | During the neoadjuvant treatment phase at baseline (week 1) and at week 13. In the adjuvant therapy phase, every 3 month, up to 12 months (from date of randomization) or date of drop out, whatever comes first
  * questions about "self care", "usual activities", "pain /discomfort", anxiety/depression" are assessed on a 5 level-scale using tick boxes : "I have no problem"; "I have slight problems"; "I have moderate problems"; "I have severe problems" "I am unable"
  * assessment of the patient health (good or bad) is measured on a scale numbered from 0 to 100 (100 means the best heath and 0 means the worst)
Health-related quality of life using EORTC QLQ-C30 scale | During the neoadjuvant treatment phase at baseline (week 1) and at week 13. In the adjuvant therapy phase, every 3 month, up to 12 months (from date of randomization) or date of drop out, whatever comes first
  * Assessment of quality of life questions (activities, breath, pain, sleep, appetite, vomiting, constipation, others..) are measured on a 4 level-scale: 1 (not at all); 2 (a little); 3 (quite a bit); 4 (very much)
  * Assessment of Overall health and overall quality of life during the past week is measured on a 7 level-scale going from 1 (very poor) to 7 (excellent)
Tumor size reduction by mammography | at screening visit and 12 weeks after start of therapy treatment
  The diameters of the tumors in the breast will be measured in millimeter by mammography as part of clinical response measure. The tumor size measurement 13 weeks after start of therapy is also used to reach a secondary endpoint: near pCR, defined as tumor sized ypT1a/is, any ypN with tumor size.
Tumor size reduction by palpation and ultrasound | at screening visit and 4, 7 and 13 weeks after start of therapy treatment
  The diameters of the tumors in the breast will be measured in millimeter by palpation and ultrasound as part of clinical response measure. The tumor size measurement 13 weeks after start of therapy is also used to reach a secondary endpoint: near pCR, defined as tumor sized ypT1a/is, any ypN with tumor size.
Overall survival | From date of randomization until the date of death from any cause, assessed up to 60 months
  The overall survival is defined as time (days) between study treatment allocation and death of patient due to any cause.
Duration of invasive disease-free survival | From date of treatment allocation until the date of first documented progression or secondary tumor or date of death from any cause, whichever came first, assessed up to 60 months (study duration including follow up)
  Duration of invasive disease-free survival is defined as time (days) between study treatment allocation and relapse, secondary tumor event or death.
Number of mastectomies | 14 weeks after start of therapy treatment
  The number of mastectomies will be determined at time of surgery (week 14 and week 18)
Ki67 level | 4 weeks after start of therapy treatment
  The level of Ki67 in biopsie material will be measured at week 4 of neoadjuvant therapy
cDNA composition | at baseline, 3 weeks, 4 weeks and 6, 18, 24, 36 48 and 60 months after start of therapy treatment
  The composition of cDNA in blood samples will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Iris Reiser, PhD, Study Director — Palleos Healthcare GmbH
Locations (1):
- Evangelisches Krankenhaus Bethesda Mönchengladbach, Mönchengladbach, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carey LA, Berry DA, Cirrincione CT, Barry WT, Pitcher BN, Harris LN, Ollila DW, Krop IE, Henry NL, Weckstein DJ, Anders CK, Singh B, Hoadley KA, Iglesia M, Cheang MC, Perou CM, Winer EP, Hudis CA. Molecular Heterogeneity and Response to Neoadjuvant Human Epidermal Growth Factor Receptor 2 Targeting in CALGB 40601, a Randomized Phase III Trial of Paclitaxel Plus Trastuzumab With or Without Lapatinib. J Clin Oncol. 2016 Feb 20;34(6):542-9. doi: 10.1200/JCO.2015.62.1268. Epub 2015 Nov 2. PMID 26527775
- [Background] Vaz-Luis I, Ottesen RA, Hughes ME, Marcom PK, Moy B, Rugo HS, Theriault RL, Wilson J, Niland JC, Weeks JC, Lin NU. Impact of hormone receptor status on patterns of recurrence and clinical outcomes among patients with human epidermal growth factor-2-positive breast cancer in the National Comprehensive Cancer Network: a prospective cohort study. Breast Cancer Res. 2012 Oct 1;14(5):R129. doi: 10.1186/bcr3324. PMID 23025714
- [Background] Prat A, Cheang MC, Galvan P, Nuciforo P, Pare L, Adamo B, Munoz M, Viladot M, Press MF, Gagnon R, Ellis C, Johnston S. Prognostic Value of Intrinsic Subtypes in Hormone Receptor-Positive Metastatic Breast Cancer Treated With Letrozole With or Without Lapatinib. JAMA Oncol. 2016 Oct 1;2(10):1287-1294. doi: 10.1001/jamaoncol.2016.0922. PMID 27281556
- [Background] Chan A, Delaloge S, Holmes FA, Moy B, Iwata H, Harvey VJ, Robert NJ, Silovski T, Gokmen E, von Minckwitz G, Ejlertsen B, Chia SKL, Mansi J, Barrios CH, Gnant M, Buyse M, Gore I, Smith J 2nd, Harker G, Masuda N, Petrakova K, Zotano AG, Iannotti N, Rodriguez G, Tassone P, Wong A, Bryce R, Ye Y, Yao B, Martin M; ExteNET Study Group. Neratinib after trastuzumab-based adjuvant therapy in patients with HER2-positive breast cancer (ExteNET): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):367-377. doi: 10.1016/S1470-2045(15)00551-3. Epub 2016 Feb 10. PMID 26874901
- [Background] Loibl S, von Minckwitz G, Blohmer J, et al: pCR as a Surrogate in HER2-Positive Patients Treated with Trastuzumab. Supplement to Cancer Research 71:[S5-4] 2011
- [Background] Tolaney SM, Barry WT, Dang CT, Yardley DA, Moy B, Marcom PK, Albain KS, Rugo HS, Ellis M, Shapira I, Wolff AC, Carey LA, Overmoyer BA, Partridge AH, Guo H, Hudis CA, Krop IE, Burstein HJ, Winer EP. Adjuvant paclitaxel and trastuzumab for node-negative, HER2-positive breast cancer. N Engl J Med. 2015 Jan 8;372(2):134-41. doi: 10.1056/NEJMoa1406281. PMID 25564897
- [Background] Harbeck N, Gluz O, Christgen M, Kates RE, Braun M, Kuemmel S, Schumacher C, Potenberg J, Kraemer S, Kleine-Tebbe A, Augustin D, Aktas B, Forstbauer H, Tio J, von Schumann R, Liedtke C, Grischke EM, Schumacher J, Wuerstlein R, Kreipe HH, Nitz UA. De-Escalation Strategies in Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Early Breast Cancer (BC): Final Analysis of the West German Study Group Adjuvant Dynamic Marker-Adjusted Personalized Therapy Trial Optimizing Risk Assessment and Therapy Response Prediction in Early BC HER2- and Hormone Receptor-Positive Phase II Randomized Trial-Efficacy, Safety, and Predictive Markers for 12 Weeks of Neoadjuvant Trastuzumab Emtansine With or Without Endocrine Therapy (ET) Versus Trastuzumab Plus ET. J Clin Oncol. 2017 Sep 10;35(26):3046-3054. doi: 10.1200/JCO.2016.71.9815. Epub 2017 Jul 6. PMID 28682681
- [Background] Gianni L, Pienkowski T, Im Y-H, et al: Five-year analysis of the phase II NeoSphere trial evaluating four cycles of neoadjuvant docetaxel (D) and/or trastuzumab (T) and/or pertuzumab (P). ASCO Meeting Abstracts 33:505, 2015
- [Background] Rimawi MF, Niravath P, Wang T, Rexer BN, Forero A, Wolff AC, Nanda R, Storniolo AM, Krop I, Goetz MP, Nangia JR, Jiralerspong S, Pavlick A, Veeraraghavan J, De Angelis C, Gutierrez C, Schiff R, Hilsenbeck SG, Osborne CK; Translational Breast Cancer Research Consortium. TBCRC023: A Randomized Phase II Neoadjuvant Trial of Lapatinib Plus Trastuzumab Without Chemotherapy for 12 versus 24 Weeks in Patients with HER2-Positive Breast Cancer. Clin Cancer Res. 2020 Feb 15;26(4):821-827. doi: 10.1158/1078-0432.CCR-19-0851. Epub 2019 Oct 29. PMID 31662331
- [Background] Gluz O, Nitz U, Liedtke C, et al: Abstract S6-07: Comparison of 12 weeks neoadjuvant Nab-paclitaxel combined with carboplatinum vs. gemcitabine in triple- negative breast cancer: WSG-ADAPT TN randomized phase II trial. Cancer Research 76:S6-07, 2016
- [Background] Francis PA, Regan MM, Fleming GF. Adjuvant ovarian suppression in premenopausal breast cancer. N Engl J Med. 2015 Apr 23;372(17):1673. doi: 10.1056/NEJMc1502618. No abstract available. PMID 25901437
- [Background] Dowsett M, Smith IE, Ebbs SR, Dixon JM, Skene A, A'Hern R, Salter J, Detre S, Hills M, Walsh G; IMPACT Trialists Group. Prognostic value of Ki67 expression after short-term presurgical endocrine therapy for primary breast cancer. J Natl Cancer Inst. 2007 Jan 17;99(2):167-70. doi: 10.1093/jnci/djk020. PMID 17228000
- [Background] Ellis MJ, Tao Y, Luo J, A'Hern R, Evans DB, Bhatnagar AS, Chaudri Ross HA, von Kameke A, Miller WR, Smith I, Eiermann W, Dowsett M. Outcome prediction for estrogen receptor-positive breast cancer based on postneoadjuvant endocrine therapy tumor characteristics. J Natl Cancer Inst. 2008 Oct 1;100(19):1380-8. doi: 10.1093/jnci/djn309. Epub 2008 Sep 23. PMID 18812550
- [Background] Ellis M, Luo J, Tao Y, et al: Tumor Ki67 Proliferation Index within 4 Weeks of Initiating Neoadjuvant Endocrine Therapy for Early Identification of Non-Responders. Cancer Res 69, 2010
- [Background] Nitz U, Gluz O, Christgen M, et al: Final analysis of WSG-ADAPT HER2+/HR- trial: Efficacy, safety, and predictive markers for 12-weeks of neoadjuvant dual blockade with trastuzumab + pertuzumab {+/-} weekly paclitaxel in HER2+/HR- early breast cancer (EBC). ASCO Meeting Abstracts 34:518, 2016
- [Background] Slamon DJ, Clark GM, Wong SG, Levin WJ, Ullrich A, McGuire WL. Human breast cancer: correlation of relapse and survival with amplification of the HER-2/neu oncogene. Science. 1987 Jan 9;235(4785):177-82. doi: 10.1126/science.3798106.
- [Background] Rouzier R, Perou CM, Symmans WF, Ibrahim N, Cristofanilli M, Anderson K, Hess KR, Stec J, Ayers M, Wagner P, Morandi P, Fan C, Rabiul I, Ross JS, Hortobagyi GN, Pusztai L. Breast cancer molecular subtypes respond differently to preoperative chemotherapy. Clin Cancer Res. 2005 Aug 15;11(16):5678-85. doi: 10.1158/1078-0432.CCR-04-2421. PMID 16115903
- [Background] Von Minckwitz G, Untch M, Nueesch E, et al: Impact of treatment characteristics on response of different breast cancer subtypes: Pooled multilayer analysis of the German neoadjuvant chemotherapy trials. J Clin Oncol (Meeting Abstracts) 28:501-, 2010
- [Background] Ellis MJ, Coop A, Singh B, Tao Y, Llombart-Cussac A, Janicke F, Mauriac L, Quebe-Fehling E, Chaudri-Ross HA, Evans DB, Miller WR. Letrozole inhibits tumor proliferation more effectively than tamoxifen independent of HER1/2 expression status. Cancer Res. 2003 Oct 1;63(19):6523-31. PMID 14559846
- [Background] Slamon DJ, Leyland-Jones B, Shak S, Fuchs H, Paton V, Bajamonde A, Fleming T, Eiermann W, Wolter J, Pegram M, Baselga J, Norton L. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med. 2001 Mar 15;344(11):783-92. doi: 10.1056/NEJM200103153441101. PMID 11248153
- [Background] Romond EH, Perez EA, Bryant J, Suman VJ, Geyer CE Jr, Davidson NE, Tan-Chiu E, Martino S, Paik S, Kaufman PA, Swain SM, Pisansky TM, Fehrenbacher L, Kutteh LA, Vogel VG, Visscher DW, Yothers G, Jenkins RB, Brown AM, Dakhil SR, Mamounas EP, Lingle WL, Klein PM, Ingle JN, Wolmark N. Trastuzumab plus adjuvant chemotherapy for operable HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1673-84. doi: 10.1056/NEJMoa052122. PMID 16236738
- [Background] Dowsett M, Allred C, Knox J, Quinn E, Salter J, Wale C, Cuzick J, Houghton J, Williams N, Mallon E, Bishop H, Ellis I, Larsimont D, Sasano H, Carder P, Cussac AL, Knox F, Speirs V, Forbes J, Buzdar A. Relationship between quantitative estrogen and progesterone receptor expression and human epidermal growth factor receptor 2 (HER-2) status with recurrence in the Arimidex, Tamoxifen, Alone or in Combination trial. J Clin Oncol. 2008 Mar 1;26(7):1059-65. doi: 10.1200/JCO.2007.12.9437. Epub 2008 Jan 28. PMID 18227529
- [Background] Kennecke H, Yerushalmi R, Woods R, Cheang MC, Voduc D, Speers CH, Nielsen TO, Gelmon K. Metastatic behavior of breast cancer subtypes. J Clin Oncol. 2010 Jul 10;28(20):3271-7. doi: 10.1200/JCO.2009.25.9820. Epub 2010 May 24. PMID 20498394
- [Background] Untch M, Gelber RD, Jackisch C, Procter M, Baselga J, Bell R, Cameron D, Bari M, Smith I, Leyland-Jones B, de Azambuja E, Wermuth P, Khasanov R, Feng-Yi F, Constantin C, Mayordomo JI, Su CH, Yu SY, Lluch A, Senkus-Konefka E, Price C, Haslbauer F, Suarez Sahui T, Srimuninnimit V, Colleoni M, Coates AS, Piccart-Gebhart MJ, Goldhirsch A; HERA Study Team. Estimating the magnitude of trastuzumab effects within patient subgroups in the HERA trial. Ann Oncol. 2008 Jun;19(6):1090-6. doi: 10.1093/annonc/mdn005. Epub 2008 Feb 21. PMID 18296421
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] Prat A, Carey LA, Adamo B, Vidal M, Tabernero J, Cortes J, Parker JS, Perou CM, Baselga J. Molecular features and survival outcomes of the intrinsic subtypes within HER2-positive breast cancer. J Natl Cancer Inst. 2014 Aug 19;106(8):dju152. doi: 10.1093/jnci/dju152. Print 2014 Aug. PMID 25139534
- [Background] Dawood S, Broglio K, Buzdar AU, Hortobagyi GN, Giordano SH. Prognosis of women with metastatic breast cancer by HER2 status and trastuzumab treatment: an institutional-based review. J Clin Oncol. 2010 Jan 1;28(1):92-8. doi: 10.1200/JCO.2008.19.9844. Epub 2009 Nov 23. PMID 19933921
- [Background] Piccart-Gebhart MJ, Procter M, Leyland-Jones B, Goldhirsch A, Untch M, Smith I, Gianni L, Baselga J, Bell R, Jackisch C, Cameron D, Dowsett M, Barrios CH, Steger G, Huang CS, Andersson M, Inbar M, Lichinitser M, Lang I, Nitz U, Iwata H, Thomssen C, Lohrisch C, Suter TM, Ruschoff J, Suto T, Greatorex V, Ward C, Straehle C, McFadden E, Dolci MS, Gelber RD; Herceptin Adjuvant (HERA) Trial Study Team. Trastuzumab after adjuvant chemotherapy in HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1659-72. doi: 10.1056/NEJMoa052306. PMID 16236737
- [Background] Joensuu H, Kellokumpu-Lehtinen PL, Bono P, Alanko T, Kataja V, Asola R, Utriainen T, Kokko R, Hemminki A, Tarkkanen M, Turpeenniemi-Hujanen T, Jyrkkio S, Flander M, Helle L, Ingalsuo S, Johansson K, Jaaskelainen AS, Pajunen M, Rauhala M, Kaleva-Kerola J, Salminen T, Leinonen M, Elomaa I, Isola J; FinHer Study Investigators. Adjuvant docetaxel or vinorelbine with or without trastuzumab for breast cancer. N Engl J Med. 2006 Feb 23;354(8):809-20. doi: 10.1056/NEJMoa053028. PMID 16495393
- [Background] Perez E, Suman V, Davidson N, et al: Results of Chemotherapy Alone, with Sequential or Concurrent Addition of 52 Weeks of Trastuzumab in the NCCTG N9831 HER2-Positive Adjuvant Breast Cancer Trial. Cancer Res 69:Abstract 80, 2010
- [Background] Swain SM, Baselga J, Kim SB, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Heeson S, Clark E, Ross G, Benyunes MC, Cortes J; CLEOPATRA Study Group. Pertuzumab, trastuzumab, and docetaxel in HER2-positive metastatic breast cancer. N Engl J Med. 2015 Feb 19;372(8):724-34. doi: 10.1056/NEJMoa1413513. PMID 25693012
- [Background] Baselga J, Cortes J, Kim SB, Im SA, Hegg R, Im YH, Roman L, Pedrini JL, Pienkowski T, Knott A, Clark E, Benyunes MC, Ross G, Swain SM; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med. 2012 Jan 12;366(2):109-19. doi: 10.1056/NEJMoa1113216. Epub 2011 Dec 7. PMID 22149875
- [Background] Geyer CE, Forster J, Lindquist D, Chan S, Romieu CG, Pienkowski T, Jagiello-Gruszfeld A, Crown J, Chan A, Kaufman B, Skarlos D, Campone M, Davidson N, Berger M, Oliva C, Rubin SD, Stein S, Cameron D. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med. 2006 Dec 28;355(26):2733-43. doi: 10.1056/NEJMoa064320. PMID 17192538
- [Background] Verma S, Miles D, Gianni L, Krop IE, Welslau M, Baselga J, Pegram M, Oh DY, Dieras V, Guardino E, Fang L, Lu MW, Olsen S, Blackwell K; EMILIA Study Group. Trastuzumab emtansine for HER2-positive advanced breast cancer. N Engl J Med. 2012 Nov 8;367(19):1783-91. doi: 10.1056/NEJMoa1209124. Epub 2012 Oct 1. PMID 23020162
- [Background] Liedtke C, Mazouni C, Hess KR, Andre F, Tordai A, Mejia JA, Symmans WF, Gonzalez-Angulo AM, Hennessy B, Green M, Cristofanilli M, Hortobagyi GN, Pusztai L. Response to neoadjuvant therapy and long-term survival in patients with triple-negative breast cancer. J Clin Oncol. 2008 Mar 10;26(8):1275-81. doi: 10.1200/JCO.2007.14.4147. Epub 2008 Feb 4. PMID 18250347
- [Background] Gianni L, Eiermann W, Semiglazov V, Manikhas A, Lluch A, Tjulandin S, Zambetti M, Vazquez F, Byakhow M, Lichinitser M, Climent MA, Ciruelos E, Ojeda B, Mansutti M, Bozhok A, Baronio R, Feyereislova A, Barton C, Valagussa P, Baselga J. Neoadjuvant chemotherapy with trastuzumab followed by adjuvant trastuzumab versus neoadjuvant chemotherapy alone, in patients with HER2-positive locally advanced breast cancer (the NOAH trial): a randomised controlled superiority trial with a parallel HER2-negative cohort. Lancet. 2010 Jan 30;375(9712):377-84. doi: 10.1016/S0140-6736(09)61964-4. PMID 20113825
- [Background] Buzdar AU, Ibrahim NK, Francis D, Booser DJ, Thomas ES, Theriault RL, Pusztai L, Green MC, Arun BK, Giordano SH, Cristofanilli M, Frye DK, Smith TL, Hunt KK, Singletary SE, Sahin AA, Ewer MS, Buchholz TA, Berry D, Hortobagyi GN. Significantly higher pathologic complete remission rate after neoadjuvant therapy with trastuzumab, paclitaxel, and epirubicin chemotherapy: results of a randomized trial in human epidermal growth factor receptor 2-positive operable breast cancer. J Clin Oncol. 2005 Jun 1;23(16):3676-85. doi: 10.1200/JCO.2005.07.032. Epub 2005 Feb 28. PMID 15738535
- [Background] Untch M, Fasching P, Konecny G, et al: Pathological Complete Response after Neoadjuvant Chemotherapy + Trastuzumab Treatment Predicts Survival and Detects a Patient Subgroup at High Need for Improvement of Anti-HER2 Therapy. Three Year Median Follow-Up Data of the TECHNO Trial. Cancer Res 71:P1-11-03, 2011
- [Background] Robidoux A, Tang G, Rastogi P, Geyer CE Jr, Azar CA, Atkins JN, Fehrenbacher L, Bear HD, Baez-Diaz L, Sarwar S, Margolese RG, Farrar WB, Brufsky AM, Shibata HR, Bandos H, Paik S, Costantino JP, Swain SM, Mamounas EP, Wolmark N. Lapatinib as a component of neoadjuvant therapy for HER2-positive operable breast cancer (NSABP protocol B-41): an open-label, randomised phase 3 trial. Lancet Oncol. 2013 Nov;14(12):1183-92. doi: 10.1016/S1470-2045(13)70411-X. Epub 2013 Oct 4. PMID 24095300
- [Background] Von Minckwitz G, Kaufmann M, Kuemmel S, et al: Correlation of various pathologic complete response (pCR) definitions with long-term outcome and the prognostic value of pCR in various breast cancer subtypes: Results from the German neoadjuvant meta-analysis. J Clin Oncol 29:abstr 1028, 2011
- [Background] Guarneri V, Broglio K, Kau SW, Cristofanilli M, Buzdar AU, Valero V, Buchholz T, Meric F, Middleton L, Hortobagyi GN, Gonzalez-Angulo AM. Prognostic value of pathologic complete response after primary chemotherapy in relation to hormone receptor status and other factors. J Clin Oncol. 2006 Mar 1;24(7):1037-44. doi: 10.1200/JCO.2005.02.6914. PMID 16505422
- [Background] de Azambuja E, Holmes AP, Piccart-Gebhart M, Holmes E, Di Cosimo S, Swaby RF, Untch M, Jackisch C, Lang I, Smith I, Boyle F, Xu B, Barrios CH, Perez EA, Azim HA Jr, Kim SB, Kuemmel S, Huang CS, Vuylsteke P, Hsieh RK, Gorbunova V, Eniu A, Dreosti L, Tavartkiladze N, Gelber RD, Eidtmann H, Baselga J. Lapatinib with trastuzumab for HER2-positive early breast cancer (NeoALTTO): survival outcomes of a randomised, open-label, multicentre, phase 3 trial and their association with pathological complete response. Lancet Oncol. 2014 Sep;15(10):1137-46. doi: 10.1016/S1470-2045(14)70320-1. Epub 2014 Aug 14. PMID 25130998
- [Background] Gianni L, Pienkowski T, Im Y-H, et al: Neoadjuvant Pertuzumab (P) and Trastuzumab (H): Antitumor and Safety Analysis of a Randomized Phase II Study ('NeoSphere'). Cancer Res 71:[S3-2], 2011
- [Background] Schneeweiss A, Chia S, Hickish T, et al: Neoadjuvant Pertuzumab and Trastuzumab Concurrent or Sequential with an Anthracycline-Containing or Concurrent with an Anthracycline-Free Standard Regimen: A Randomized Phase II Study (TRYPHAENA). Supplement to Cancer Research 71:[S5-6] 2011
- [Background] Hurvitz SA, Martin M, Symmans WF, et al: Pathologic complete response (pCR) rates after neoadjuvant trastuzumab emtansine (T-DM1 [K]) + pertuzumab (P) vs docetaxel + carboplatin + trastuzumab + P (TCHP) treatment in patients with HER2-positive (HER2+) early breast cancer (EBC) (KRISTINE). ASCO Meeting Abstracts 34:500, 2016
- [Background] Loi S, Dafni U, Karlis D, Polydoropoulou V, Young BM, Willis S, Long B, de Azambuja E, Sotiriou C, Viale G, Ruschoff J, Piccart MJ, Dowsett M, Michiels S, Leyland-Jones B. Effects of Estrogen Receptor and Human Epidermal Growth Factor Receptor-2 Levels on the Efficacy of Trastuzumab: A Secondary Analysis of the HERA Trial. JAMA Oncol. 2016 Aug 1;2(8):1040-7. doi: 10.1001/jamaoncol.2016.0339. PMID 27100299
- [Background] Piccart-Gebhart M, Holmes E, Baselga J, de Azambuja E, Dueck AC, Viale G, Zujewski JA, Goldhirsch A, Armour A, Pritchard KI, McCullough AE, Dolci S, McFadden E, Holmes AP, Tonghua L, Eidtmann H, Dinh P, Di Cosimo S, Harbeck N, Tjulandin S, Im YH, Huang CS, Dieras V, Hillman DW, Wolff AC, Jackisch C, Lang I, Untch M, Smith I, Boyle F, Xu B, Gomez H, Suter T, Gelber RD, Perez EA. Adjuvant Lapatinib and Trastuzumab for Early Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer: Results From the Randomized Phase III Adjuvant Lapatinib and/or Trastuzumab Treatment Optimization Trial. J Clin Oncol. 2016 Apr 1;34(10):1034-42. doi: 10.1200/JCO.2015.62.1797. Epub 2015 Nov 23. PMID 26598744
- [Background] Rimawi MF, Mayer IA, Forero A, Nanda R, Goetz MP, Rodriguez AA, Pavlick AC, Wang T, Hilsenbeck SG, Gutierrez C, Schiff R, Osborne CK, Chang JC. Multicenter phase II study of neoadjuvant lapatinib and trastuzumab with hormonal therapy and without chemotherapy in patients with human epidermal growth factor receptor 2-overexpressing breast cancer: TBCRC 006. J Clin Oncol. 2013 May 10;31(14):1726-31. doi: 10.1200/JCO.2012.44.8027. Epub 2013 Apr 8. PMID 23569315
- [Background] Guarneri V, Chavez-Mac Gregor M, Hsu L, et al: Use of Ki-67 in residual disease following preoperative chemotherapy to predict of recurrence and death in breast cancer patients. J Clin Oncol (Meeting Abstracts) 28:621-, 2010
- [Background] Giuliano AE, Hunt KK, Ballman KV, Beitsch PD, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, McCall LM, Morrow M. Axillary dissection vs no axillary dissection in women with invasive breast cancer and sentinel node metastasis: a randomized clinical trial. JAMA. 2011 Feb 9;305(6):569-75. doi: 10.1001/jama.2011.90. PMID 21304082
- [Background] Whelan TJ, Olivotto I, Ackerman I, et al: NCIC-CTG MA.20: An intergroup trial of regional nodal irradiation in early breast cancer. J Clin Oncol Suppl:LBA1003, 2011
- [Background] Marinovich ML, Houssami N, Macaskill P, von Minckwitz G, Blohmer JU, Irwig L. Accuracy of ultrasound for predicting pathologic response during neoadjuvant therapy for breast cancer. Int J Cancer. 2015 Jun 1;136(11):2730-7. doi: 10.1002/ijc.29323. Epub 2014 Nov 25. PMID 25387885
- [Background] Gourgou-Bourgade S, Cameron D, Poortmans P, Asselain B, Azria D, Cardoso F, A'Hern R, Bliss J, Bogaerts J, Bonnefoi H, Brain E, Cardoso MJ, Chibaudel B, Coleman R, Cufer T, Dal Lago L, Dalenc F, De Azambuja E, Debled M, Delaloge S, Filleron T, Gligorov J, Gutowski M, Jacot W, Kirkove C, MacGrogan G, Michiels S, Negreiros I, Offersen BV, Penault Llorca F, Pruneri G, Roche H, Russell NS, Schmitt F, Servent V, Thurlimann B, Untch M, van der Hage JA, van Tienhoven G, Wildiers H, Yarnold J, Bonnetain F, Mathoulin-Pelissier S, Bellera C, Dabakuyo-Yonli TS. Guidelines for time-to-event end point definitions in breast cancer trials: results of the DATECAN initiative (Definition for the Assessment of Time-to-event Endpoints in CANcer trials)dagger. Ann Oncol. 2015 May;26(5):873-879. doi: 10.1093/annonc/mdv106. Epub 2015 Feb 27. PMID 25725046
- [Derived] Gluz O, Nitz UA, Christgen M, Kuemmel S, Holtschmidt J, Schumacher J, Hartkopf A, Potenberg J, Luedtke-Heckenkamp K, Just M, Schem C, von Schumann R, Kolberg-Liedtke C, Eulenburg CZ, Schinkothe T, Graeser M, Wuerstlein R, Kates RE, Kreipe HH, Harbeck N. Efficacy of Endocrine Therapy Plus Trastuzumab and Pertuzumab vs De-escalated Chemotherapy in Patients with Hormone Receptor-Positive/ERBB2-Positive Early Breast Cancer: The Neoadjuvant WSG-TP-II Randomized Clinical Trial. JAMA Oncol. 2023 Jul 1;9(7):946-954. doi: 10.1001/jamaoncol.2023.0646. PMID 37166817